CLINICAL TRIAL: NCT06299033
Title: A Phase 1 Dose-escalation, Single-Center, Open-labeled Study to Evaluate the Safety and Tolerability of Human Induced Pluripotent Stem Cell-derived Human Forebrain Neural Progenitor Cell Injection (hNPC01) in Chronic Ischemic Stroke
Brief Title: A Safety and Tolerability Study of Human Forebrain Neural Progenitor Cells Injection (hNPC01) in Subjects With Chronic Ischemic Stroke
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hopstem Biotechnology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HPS-NP1-101
Record Dates: First submitted 2024-01-27; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Chronic Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- hNPC01 therapy (Experimental): 1.5×10^7 hNPC01 cells; 3.0×10^7 hNPC01 cells; 6.0×10^7 hNPC01 cells
  Interventions: Drug: hNPC01

INTERVENTIONS:
Drug: hNPC01 — hNPC01, human forebrain neural progenitor cell product, intracerebral injection

SUMMARY:
The principal aims of the clinical investigation involve assessing the safety profile and MTD of human forebrain neural progenitor cells (hNPC01) administered at escalated doses via single-dose intracerebral injection to subjects with stable chronic ischemic stroke.

DETAILED DESCRIPTION:
The primary aims of this open-label single-armed study is to evaluate the safety and tolerability up to 4 cohorts of escalating doses of hNPC01 administered at a single dose via intracerebral injection to subjects with chronic cerebral ischemic stroke, and to determine MTD. The exploratory aim is to explore the evaluation tools with preliminary efficacy assessment and the potential of hNPC01 to mitigate the symptoms, especially motor symptoms associated with chronic stroke. Eligible participants for this study are individuals who have experienced a single ischemic stroke 6 to 60 months prior of enrollment and have exhibited no significant improvement following standard physical therapy interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or his/her legal guardian must understand and voluntarily sign an Informed Consent Form (ICF) prior to any study-related assessments/procedure being conducted;
2. Age 30-65 years old, male or female; at the time of signing the ICF;
3. Female patients with negative blood pregnancy test and women in the reproductive period need to adopt effective contraceptive methods; Or has become infertile (menopausal for at least 2 years or has undergone hysterectomy, oophorectomy, or sterilization surgery); Male patients who have no plans to donate sperm or have children within 30 days before the trial and six months after the trial end need to adopt effective contraceptive methods;
4. Documented history of completed ischemic stroke in the subcortical and/or cortical regions of the middle cerebral artery (MCA) or lenticulostriate arteries confirmed by head CT or magnetic resonance imaging;
5. 6 - 60 months since the acute onset of ischemic stroke, accompanied by unilateral limb motor dysfunction, with/without aphasia;
6. Modified Rankin Score 3, or 4 points at time of screening;
7. FMMS scores lower than 55 and score changes no greater than 5 points in two assessments at least 3 weeks apart before surgery;
8. NIHSS score change is no greater than 4 points in two assessments at least 3 weeks apart before surgery;
9. Subject must have maintained regular physical therapy and rehabilitation prior to enrollment and be able to continue physical therapy and rehabilitation after treatment.

Exclusion Criteria:

1. Has any psychological or psychiatric condition that would significantly interfere with the study;
2. History of more than one symptomatic stroke [transient ischemic attacks (TIAs) are not exclusionary];
3. Has signs and symptoms of intracerebral hernia or elevated intracerebral pressure;
4. History of epilepsy or current use of antiepileptic drugs, including any seizures in the 3 months prior to screening;
5. Intracerebral aneurysm or arteriovenous malformation; hemorrhagic transformation of ischemic loci within 2 weeks of screening; moyamoya disease (MMD); autosomal dominant cerebrovascular disease with subcortical infarction and leukoencephalopathy; patients with giant cerebral infarction (MRI confirms that the infarct size is greater than 150 cm^3); CT angiography (CTA) shows severe stenosis in vital vessels in head or neck;
6. Patients with severely impaired motor function of one limb caused by previous neurological diseases (such as PD, motor neuron disease, arthritis, or anatomical deformity, etc.); Patients who have undergone any major surgery 8 weeks prior to screening;
7. Severe muscular atrophy or muscular dystrophy;
8. Patients with severe cardiovascular diseases within 3 months of screening, such as malignant arrhythmia, atrial fibrillation, acute myocardial infarction, congestive heart failure, etc. (cardiac function grade III-IV using the New York Heart Association (NYHA) classification for heart failure);
9. Patients participating in other drug or device clinical trials within the last 3 months or 5 half-lives of the drug, whichever is longer;
10. Receiving other cell transfusions or alike other than transfusion in the past 5 years;
11. Any of the following diseases or conditions:

    1. Severe coagulopathy, preoperative INR (International Normalized Ratio)>1.4;
    2. Patients with positive HLA (Human Leukocyte Antigen) before surgery;
    3. Severe active infection with poor drug control before surgery;
    4. Severe dermatitis or severe skin damage in the operation area;
    5. History of tumors other than benign tumors; history of brain tumors, including meningiomas;
    6. Laboratory values meeting any of the following criteria (a second retest can be performed for patients with a first test result outside the specified range, and the patients can be included in the study if the second test results are evaluated by the investigator as normal):

       * Hemoglobin <90 g/L
       * White blood cell count (WBC)<3.5×10^9/L
       * Neutrophil count <1.5×10^9/L
       * Platelet count <100×10^9/L
       * Serum alanine aminotransferase (ALT), aspartate aminotransferase (AST) 2 times the upper limit of normal (ULN)
       * Serum creatinine >1.2 × ULN
    7. Uncontrolled or poorly controlled hypertension despite medicine (systolic blood pressure >160 mmHg, or diastolic blood pressure >100 mmHg) or hypotension requiring pressor therapy;
    8. Uncontrolled or poorly controlled diabetes despite medicine (glycosylated hemoglobin A1c > 8%);
    9. Active gastrointestinal bleeding;
    10. Positive active pulmonary tuberculosis (if positive γ-interferon release test in screening period and the safety risk is within a controllable range after evaluation by the investigators, the participant can be enrolled);
    11. Active hepatitis B patients, including positive Hepatitis B surface antigens (HBsAg), and patients who had hepatitis B virus (HBV) infection in the past and whose HBV infection has disappeared (defined as hepatitis B core antibody [HBcAb] positive and HBsAg negative) meet the inclusion criteria;
    12. Hepatitis C virus antibody positive;
    13. Syphilis infected subjects (subjects who test positive for Treponema pallidum serology need to undergo further non-Treponema pallidum serology tests. If the test result is negative, the investigators determine that patients who have previously been infected with syphilis but have recovered meet the inclusion criteria);
    14. HIV antibody positive
12. Primary or secondary immunodeficiency; or any medical condition involving immunosuppressants intake;
13. Persistent MRI artifacts, no clear MRI images can be obtained before or after surgery; patients with contraindications to MRI or PET scans;
14. Contraindications to cyclosporine or methylprednisone sodium succinate or prednisone;
15. Neither able or willing to participate in physical and/or professional therapy as scheduled, nor to return to the hospital on time for follow-up visits as planned;
16. Inability to discontinue antiplatelet or anticoagulant medications within the perioperative period;
17. Existence of recent drug abuse or alcohol abuse or any other medical conditions that, in the opinion of the investigator, could interfere with the clinical study results or compromise the clinical condition of the subject, or which in the opinion of the investigator, could increase procedural complications.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by physiological parameters during 6 months after intracerebral injection of hNPC01 | during 6 months after intracerebral hNPC01 injection

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by physiological parameters during 12 months after intracerebral injection of hNPC01 | during 12 months after intracerebral hNPC01 injection

OTHER OUTCOMES:
Number of participants with motor function improvement as assessed by rating scales of Modified Rankin Scale (mRS) during 12 months of treatment | during 12 months after intracerebral hNPC01 injection
  mRS ranges from 0~6 points, higher scores mean a worse outcome
Number of participants with motor function improvement as assessed by rating scales of Fugl-Meyer Motor Scale (FMMS) during 12 months of treatment | during 12 months after intracerebral hNPC01 injection
  FMMS ranges from 0~100 points, higher scores mean a better outcome
Number of participants with motor function improvement as assessed by rating scales of NIH Stroke Scale (NIHSS) during 12 months of treatment | during 12 months after intracerebral hNPC01 injection
  NIHSS ranges from 0~42 points, higher scores mean a worse outcome
Number of participants with motor function improvement as assessed by rating scales of Barthel Index (BI) during 12 months of treatment | during 12 months after intracerebral hNPC01 injection
  BI ranges from 0~100 points, higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- XiangYa Hospital, Changsha, Hunan, China